CLINICAL TRIAL: NCT00734071
Title: A Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Fixed-Dose Study Comparing the Efficacy and Safety of Single Dose of Lu AA21004 in Acute Treatment of Adults With Generalized Anxiety Disorder
Brief Title: An Efficacy and Safety Study of Vortioxetine (Lu AA21004) in Treating Generalized Anxiety Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LuAA21004_310; U1111-1114-4876 (Registry Identifier: WHO)
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Results first posted 2013-12-18 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-10

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized Anxiety Disorder; Mood Disorder; Affective Disorder; Anxiety Disorder; Drug Therapy
MeSH Terms: conditions — Generalized Anxiety Disorder; Mood Disorders; Anxiety Disorders | interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Vortioxetine placebo-matching capsules, orally, once daily for up to 8 weeks.
  Interventions: Drug: Placebo
- Vortioxetine 5 mg (Experimental): Vortioxetine 5 mg, encapsulated tablets, orally, once daily for up to 8 weeks.
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — Encapsulated vortioxetine immediate-release tablets
  Other Names: Lu AA21004; Brintellix®
  Arms: Vortioxetine 5 mg
Drug: Placebo — Vortioxetine placebo-matching capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and efficacy of vortioxetine, once daily (QD), in treating Generalized Anxiety Disorder.

DETAILED DESCRIPTION:
The drug that was tested in this study is called Vortioxetine. Vortioxetine is being tested to treat anxiety in adults who have general anxiety disorder (GAD). This study looked at GAD relief in people who took vortioxetine.

The study enrolled 304 patients. Participants were randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which remained undisclosed to the patient and study doctor during the study (unless there was an urgent medical need):

* Vortioxetine 5 mg
* Placebo (dummy inactive pill) - this was a capsule that looked like the study drug but had no active ingredient.

All participants were asked to take one capsule at the same time each day throughout the study.

This multi-center trial was conducted in the United States. The overall time to participate in this study was up to 13 weeks. Participants made 7 visits to the clinic, and were contacted by telephone 4 weeks after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Has a primary diagnosis of Generalized Anxiety Disorder according to the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR®) criteria.
* Has a Hamilton Anxiety Scale total score greater than or equal to 20 at Screening and Baseline.
* Has a Hamilton Anxiety Scale score greater than or equal to 2 on both Item 1 (anxious mood) and Item 2 (tension) at Screening and Baseline.
* Has a Montgomery-Åsberg Depression Rating Scale total score less than or equal to 16 at Screening and Baseline.

Exclusion Criteria:

* Has 1 or more of the following:

  * Any current psychiatric disorder other than Generalized Anxiety Disorder as defined in the DSM-IV-TR (as assessed by the Mini International Neuropsychiatric Interview [MINI]).
  * Current or past history of: manic or hypomanic episode, schizophrenia or any other psychotic disorder, including major depression with psychotic features, mental retardation, organic mental disorders, or mental disorders due to a general medical condition as defined in the DSM-IV-TR.
  * Any substance disorder (except nicotine and caffeine) within the previous 6 months as defined in the DSM-IV-TR® and subject must have a negative urine drug screen prior to Baseline.
  * Presence or history of a clinically significant neurological disorder (including epilepsy).
  * Neurodegenerative disorder (Alzheimer disease, Parkinson disease, multiple sclerosis, Huntington disease, etc.).
  * Any Axis II disorder that might compromise the study.
* Is taking excluded medications.
* Has a significant risk of suicide according to the investigator's opinion or has a score greater than or equal to 5 on Item 10 (suicidal thoughts) of the Montgomery-Åsberg Depression Rating Scale or has made a suicide attempt in the previous 6 months.
* Has previously failed to respond to adequate treatment with selective serotonin reuptake inhibitors and/or serotonin-norepinephrine reuptake inhibitors.
* Has received electroconvulsive therapy within 6 months prior to Screening.
* Is currently receiving formal cognitive or behavioral therapy, systematic psychotherapy, or plans to initiate such therapy during the study.
* Has a clinically significant unstable illness.
* Has an alanine aminotransferase, aspartate aminotransferase, or total bilirubin level greater than 1.5 times the upper limit of normal.
* Has a serum creatinine of greater than 1.5 times the upper limit of normal.
* Has a previous history of cancer that had been in remission for less than 5 years.
* Has thyroid stimulating hormone value outside the normal range at Screening and is deemed clinically significant by the investigator.
* Has an abnormal electrocardiogram.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2008-06; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Clinical Science, Study Director — Takeda
Locations (33):
- United States (33):
  - Anaheim, California
  - Arcadia, California
  - Irvine, California
  - National City, California
  - Sherman Oaks, California
  - Upland, California
  - Washington D.C., District of Columbia
  - Bradenton, Florida
  - Coral Gables, Florida
  - North Miami, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Oak Brook, Illinois
  - Park Ridge, Illinois
  - Lafayette, Indiana
  - Wichita, Kansas
  - Baltimore, Maryland
  - Fall River, Massachusetts
  - Worcester, Massachusetts
  - Flowood, Mississippi
  - Brooklyn, New York
  - New York, New York
  - The Bronx, New York
  - Morganton, North Carolina
  - Cincinnati, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Lincoln, Rhode Island
  - Memphis, Tennessee
  - Austin, Texas
  - San Antonio, Texas
  - Charleston, West Virginia

REFERENCES:
- [Result] Rothschild AJ, Mahableshwarkar AR, Jacobsen P, Yan M, Sheehan DV. Vortioxetine (Lu AA21004) 5 mg in generalized anxiety disorder: results of an 8-week randomized, double-blind, placebo-controlled clinical trial in the United States. Eur Neuropsychopharmacol. 2012 Dec;22(12):858-66. doi: 10.1016/j.euroneuro.2012.07.011. Epub 2012 Aug 15. PMID 22901736

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 33 investigative sites in the United States from 25 June 2008 to 06 March 2009.
Pre-assignment Details: Participants with a diagnosis of generalized anxiety disorder were enrolled equally in one of two treatment groups, once a day placebo or 5 mg vortioxetine.
Period: Overall Study
Arm/Group | Placebo | Vortioxetine 5 mg
Started | 152 | 152
Treated | 151 | 148
Completed | 114 | 125
Not Completed | 38 | 27
Not completed — Adverse Event | 4 | 3
Not completed — Lack of Efficacy | 3 | 1
Not completed — Noncompliance | 2 | 2
Not completed — Protocol Deviations | 3 | 4
Not completed — Voluntary Withdrawal | 9 | 7
Not completed — Lost to Follow-up | 16 | 8
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vortioxetine 5 mg | Total
Number analyzed (Participants) | 152 | 152 | 304
Age Continuous [Mean (Standard Deviation); unit: years] | 41.4 (12.81) | 41.0 (14.05) | 41.2 (13.42)
Age, Customized [Number; unit: participants]
  ≤55 years | 128 | 129 | 257
  >55 years | 24 | 23 | 47
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 103 | 200
  Male | 55 | 49 | 104
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian (White, including Hispanic) | 131 | 123 | 254
  Black | 17 | 24 | 41
  Asian | 2 | 3 | 5
  American Indian or Alaska Native | 0 | 2 | 2
  Native Hawaiian/ Other Pacific Islander | 2 | 0 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 24 | 26 | 50
  Non-Hispanic/Non-Latino | 128 | 126 | 254
Region of Enrollment [Number; unit: participants]
  United States | 152 | 152 | 304
Weight [Mean (Standard Deviation); unit: kg] | 83.68 (20.916) | 80.10 (20.296) | 81.89 (20.652)
Height [Mean (Standard Deviation); unit: cm] | 167.73 (8.765) | 167.72 (9.158) | 167.73 (8.949)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.66 (6.861) | 28.42 (6.680) | 29.04 (6.789)
Smoking Classification [Number; unit: participants]
  Never Smoked | 78 | 76 | 154
  Current Smoker | 38 | 43 | 81
  Ex-smoker | 36 | 33 | 69
Alcohol Consumption [Number; unit: participants]
  Never | 48 | 39 | 87
  Once monthly or less often | 57 | 55 | 112
  Once a week | 17 | 28 | 45
  2 to 6 times per week | 27 | 27 | 54
  Daily | 3 | 3 | 6
Hamilton Anxiety Scale Total Score [Mean (Standard Deviation); unit: scores on a scale] — Hamilton Anxiety Scale (HAM-A) is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 (absent) to 56 (maximum severity).
  scores on a scale | 24.6 (3.60) | 24.7 (3.79) | 24.7 (3.69)
Clinical Global Impression - Severity scale score [Mean (Standard Deviation); unit: scores on a scale] — The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale where the clinician rates the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis on the following scale: 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill. The number of participants with available data were 151 and 152 in each treatment arm respectively.
  scores on a scale | 4.3 (0.49) | 4.3 (0.53) | 4.3 (0.51)
Hospital Anxiety and Depression - Anxiety subscale [Mean (Standard Deviation); unit: scores on a scale] — Hospital Anxiety and Depression (HAD) Anxiety sub-scale consists of 7 items that are assessed on a scale from 0 (no anxiety) to 3 (severe feeling of anxiety). The anxiety subscale determines a state of generalized anxiety including anxious mood, restlessness, anxious thoughts and panic attacks. Scores are summed and range from 0 to 21 (maximal severity). The number of participants with available data were 149 and 151 in each treatment arm respectively.
  scores on a scale | 13.5 (3.14) | 13.8 (3.39) | 13.7 (3.26)
Hospital Anxiety and Depression - Depression subscale [Mean (Standard Deviation); unit: scores on a scale] — Hospital Anxiety and Depression (HAD) Depression sub-scale consists of 7 items that are assessed on a scale from 0 (no depression) to 3 (severe feeling of depression). The depression subscale focuses on the state of lost interest and diminished pleasure response. Scores are summed and range from 0 to 21 (maximal severity). The number of participants with available data were 149 and 151 in each treatment arm respectively.
  scores on a scale | 8.5 (3.79) | 8.1 (3.91) | 8.3 (3.85)
Montgomery Åsberg Depression Rating Scale (MADRS) total score [Mean (Standard Deviation); unit: scores on a scale] — The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 to 6. The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression).
  scores on a scale | 11.83 (3.007) | 12.09 (2.902) | 11.96 (2.953)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Hamilton Anxiety Scale (HAM-A) Total Score at Week 8
Description: The HAM-A is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 to 56 where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. Total scores above 30 are rare, but indicate very severe anxiety. Least Squares (LS) means were from a mixed model for repeated measurements (MMRM).
Time Frame: Baseline to Week 8
Population: The Full Analysis Set included all patients who were randomized, received at least 1 dose of study drug, and had at least 1 post-baseline value for assessment of primary efficacy. A mixed model for repeated measurements (MMRM) based on observed cases was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 113 | 124
scores on a scale | -13.16 (0.655) | -12.57 (0.646)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; P-values were tested at the 5% level of significance (ie, statistical significance if P<0.05). To control for multiplicity, a pre-specified sequential testing procedure was applied to compare 5 mg vortioxetine to placebo; as soon as an endpoint was non-significant at 0.05, the testing procedure stopped for all subsequent endpoints; Test type: Superiority or Other; p = 0.518, Mixed model for repeated measurements — Pre-specified sequential statistical testing procedure indicates that when p-value >0.05, hierarchical testing stops and for subsequent endpoints in the sequence a nominal p-value is provided; LS Mean Difference = 0.59, 95% CI 2-sided [-1.20 to 2.38], Standard Error of Mean 0.911

2. Secondary Outcome: Change From Baseline in the Hospital Anxiety and Depression (HAD) Anxiety Subscale at Week 8
Description: The Hospital Anxiety and Depression (HAD) Anxiety sub-scale consists of 7 items that are assessed by a scale from 0 (no anxiety) to 3 (severe feeling of anxiety). The anxiety subscale determines a state of generalized anxiety including anxious mood, restlessness, anxious thoughts and panic attacks. Scores are summed and range from 0 to 21 (maximal severity). LS means were from a mixed model for repeated measurements (MMRM).
Time Frame: Baseline to Week 8
Population: The Full Analysis Set. A mixed model for repeated measurements (MMRM) based on observed cases was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 111 | 124
scores on a scale | -4.84 (0.392) | -5.06 (0.384)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Statistical tests were 2-sided and results were presented with 95% confidence intervals with the estimated P-values at the 5% level of significance (ie, statistical significance if P<0.05); Test type: Superiority or Other; p = 0.685, Mixed model for repeated measurements — Hierarchical testing stopped at the primary endpoint in the testing sequence, a nominal p-value is provided; LS Mean Difference = -0.22, 95% CI 2-sided [-1.29 to 0.85], Standard Error of Mean 0.542

3. Secondary Outcome: Clinical Global Impression Scale-Global Improvement at Week 8
Description: The Clinical Global Impression - Global Improvement scale assesses the participant's improvement (or worsening) as assessed by the clinician relative to Baseline on a 7-point scale: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse. LS means were from a mixed model for repeated measurements (MMRM).
Time Frame: Baseline to Week 8
Population: Full analysis set. A mixed model for repeated measurements (MMRM) based on observed cases was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 113 | 124
scores on a scale | 2.25 (0.101) | 2.25 (0.099)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.984, Mixed model for repeated measurements — Statistical tests were 2-sided and results were presented with 95% confidence intervals with the estimated P-values at the 5% level of significance (ie, statistical significance if P<0.05). No adjustments for multiplicity were made; LS Mean Difference = 0.00, 95% CI 2-sided [-0.27 to 0.28], Standard Error of Mean 0.141

4. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Score at Week 8
Description: The Sheehan Disability Scale assesses functional impairment in 3 domains: work/school, social life or leisure activities, and home life or family responsibilities. The participant rates the extent to which each aspect is impaired on a 10-point visual analog scale, from 0 (not at all) to 10 (extremely). The 3 scores are added together to calculate the total score, which ranges from 0 to 30, with higher scores indicating more impairment. LS means were from a mixed model for repeated measurements (MMRM).
Time Frame: Baseline to Week 8
Population: Full analysis set. A mixed model for repeated measurements (MMRM) based on observed cases was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 91 | 97
scores on a scale | -6.68 (0.618) | -6.35 (0.616)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.703, Mixed model for repeated measurements — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = 0.33, 95% CI 2-sided [-1.38 to 2.04], Standard Error of Mean 0.866

5. Secondary Outcome: Percentage of Responders in HAM-A Total Score at Week 8
Description: Response was defined as participants with a ≥50% decrease from Baseline in the Hamilton Anxiety Scale (HAM-A) total score. The HAM-A is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 (symptoms absent) to 56 (maximum severity).
Time Frame: Baseline and Week 8
Population: Full analysis set; Last observation carried forward was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 144 | 145
percentage of participants | 50.0 | 53.1
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.602, Regression, Logistic; Logistic regression with explanatory variables for treatment and Baseline HAM-A score; Odds Ratio (OR) = 1.131, 95% CI 2-sided [0.713 to 1.795]

6. Secondary Outcome: Change From Baseline in the Hamilton Anxiety Scale (HAM-A) Total Score at Week 8 in Participants With Baseline HAM-A ≥25
Description: as for outcome 1
Time Frame: Baseline to Week 8
Population: Full analysis set patients with a HAM-A Baseline score ≥25. A mixed model for repeated measurements (MMRM) based on observed cases was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 59 | 63
scores on a scale | -14.04 (1.104) | -14.05 (1.080)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.995, Mixed model for repeated measurements — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -0.01, 95% CI 2-sided [-3.09 to 3.07], Standard Error of Mean 1.558

7. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Social Functioning Subscore at Week 8
Description: The Medical Outcomes Study SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The social functioning subscale assesses limitations in social activities because of physical or emotional problems. The sub-score scale ranges from 0 (best) - 100 (worst). LS means were from a mixed model for repeated measurements (MMRM).
Time Frame: Baseline to Week 8
Population: The Full Analysis Set. A mixed model for repeated measurements (MMRM) based on observed cases was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 113 | 125
scores on a scale | 17.43 (2.133) | 18.44 (2.091)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.731, Mixed model for repeated measurements — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = 1.02, 95% CI 2-sided [-4.79 to 6.83], Standard Error of Mean 2.951

8. Secondary Outcome: Change From Baseline in Hamilton Anxiety Scale (HAM-A) Total Score at Other Weeks Assessed
Description: as for outcome 1
Time Frame: Baseline to Weeks 1, 2, 4 and 6.
Population: The Full Analysis Set. A mixed model for repeated measurements (MMRM) based on observed cases was used. "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 144 | 145
scores on a scale
  Week 1 (n=141, 144) | -4.84 (0.415) | -4.59 (0.422)
  Week 2 (n=134, 142) | -7.78 (0.542) | -8.22 (0.541)
  Week 4 (n=131, 135) | -10.13 (0.590) | -9.82 (0.590)
  Week 6 (n=124, 129) | -12.39 (0.632) | -11.61 (0.630)

9. Secondary Outcome: Change From Baseline in the Hospital Anxiety and Depression (HAD) Anxiety Subscale at Other Weeks Assessed
Description: as for outcome 2
Time Frame: Baseline to Weeks 1 and 4
Population: The Full Analysis Set with available data at Baseline. A mixed model for repeated measurements (MMRM) based on observed cases was used; "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 140 | 144
scores on a scale
  Week 1 (n=139, 142) | -1.81 (0.269) | -2.07 (0.273)
  Week 4 (n=130, 135) | -3.41 (0.328) | -3.72 (0.329)

10. Secondary Outcome: Clinical Global Impression Scale-Global Improvement at Other Weeks Assessed
Description: as for outcome 3
Time Frame: Baseline to Weeks 1, 2, 4 and 6
Population: Full analysis set. A mixed model for repeated measurements (MMRM) based on observed cases was used; "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 144 | 145
scores on a scale
  Week 1 (n=141, 144) | 3.32 (0.066) | 3.38 (0.066)
  Week 2 (n=134, 142) | 2.92 (0.081) | 2.83 (0.081)
  Week 4 (n=131, 135) | 2.57 (0.089) | 2.57 (0.089)
  Week 6 (n=124, 129) | 2.42 (0.096) | 2.39 (0.095)

11. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Score at Other Weeks Assessed
Description: The Sheehan Disability Scale assesses functional impairment in 3 domains: work/school, social life or leisure activities, and home life or family responsibilities. The participant rates the extent to which each aspect is impaired on a 10-point visual analog scale, from 0 (not at all) to 10 (extremely). The 3 scores are added together to calculate the total score, which ranges from 0 to 30, with higher scores indicating more impairment. LS means and P-values were from a mixed model for repeated measurements (MMRM).
Time Frame: Baseline to Weeks 1, 2 and 4
Population: Full analysis set with available data at Baseline. A mixed model for repeated measurements (MMRM) based on observed cases was used; "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 124 | 121
scores on a scale
  Week 1 (n=117, 116) | -2.13 (0.484) | -2.46 (0.497)
  Week 2 (n=109, 114) | -4.35 (0.566) | -4.02 (0.572)
  Week 4 (n=106, 108) | -5.57 (0.587) | -5.38 (0.593)

12. Secondary Outcome: Percentage of Responders in HAM-A Total Score at Other Weeks Assessed
Description: as for outcome 5
Time Frame: Baseline and Weeks 1, 2, 4 and 6
Population: Full analysis set; Last observation carried forward was used; "n" indicates the number of patients included in the analysis at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 144 | 145
percentage of participants
  Week 1 (n=141, 144) | 9.9 | 6.9
  Week 2 (n=144, 145) | 22.9 | 24.1
  Week 4 (n=144, 145) | 34.7 | 37.2
  Week 6 (n=144, 145) | 47.2 | 45.5

13. Secondary Outcome: Change From Baseline in the Hamilton Anxiety Scale (HAM-A) Total Score at Other Weeks Assessed in Participants With Baseline HAM-A ≥25
Description: as for outcome 1
Time Frame: Baseline to Weeks 1, 2, 4 and 6
Population: Full analysis set patients with a HAM-A Baseline score ≥25. A mixed model for repeated measurements (MMRM) based on observed cases was used; "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 73 | 71
scores on a scale
  Week 1 (n=71, 71) | -5.39 (0.675) | -4.73 (0.648)
  Week 2 (n=70, 70) | -8.37 (0.889) | -8.94 (0.873)
  Week 4 (n=67, 67) | -10.90 (0.994) | -10.74 (0.980)
  Week 6 (n=63, 65) | -13.60 (1.040) | -12.82 (1.021)

14. Secondary Outcome: Percentage of Participants in HAM-A Remission at Each Week Assessed
Description: Remission is defined as a Hamilton Anxiety Scale (HAM-A) total score ≤ 7. The HAM-A is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 (symptoms absent) to 56 (maximum severity).
Time Frame: Weeks 1, 2, 4, 6 and 8
Population: Full analysis set; Last observation carried forward was used. "n" indicates the number of patients included in the analysis at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 144 | 145
percentage of participants
  Week 1 (n-141, 144) | 2.1 | 0.7
  Week 2 (n=144, 145) | 5.6 | 7.6
  Week 4 (n=144, 145) | 15.3 | 12.4
  Week 6 (n=144, 145) | 22.2 | 22.1
  Week 8 (n=144, 145) | 22.2 | 25.5

15. Secondary Outcome: Change From Baseline in Clinical Global Impression Scale-Severity of Illness at Each Week Assessed
Description: The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness on the following scale: 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill. LS means were from a mixed model for repeated measurements (MMRM).
Time Frame: Baseline to Weeks 1, 2, 4, 6 and 8
Population: Full analysis set. A mixed model for repeated measurements (MMRM) based on observed cases was used. "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 144 | 145
scores on a scale
  Week 1 (n=141, 144) | -0.37 (0.057) | -0.38 (0.058)
  Week 2 (n=134, 142) | -0.75 (0.081) | -0.86 (0.081)
  Week 4 (n=131, 135) | -1.15 (0.093) | -1.05 (0.092)
  Week 6 (n=124, 129) | -1.45 (0.098) | -1.40 (0.097)
  Week 8 (n=113, 124) | -1.72 (0.104) | -1.54 (0.102)

16. Secondary Outcome: Change From Baseline in the Hospital Anxiety and Depression (HAD) Depression Subscale at Each Week Assessed
Description: The HAD-Depression subscale is completed by the participant and measures depression, focusing on the state of lost interest and diminished pleasure response. The subscale is made up of 7 items that are assessed on a scale from 0 (no depression) to 3 (severe feeling of depression). Participants are required to indicate the response which most accurately reflects the way they have felt over the last few days. The item scores are summed and the total subscore ranges from 0 to 21 (maximal severity). LS means were from a mixed model for repeated measurements (MMRM).
Time Frame: Baseline to Weeks 1, 4 and 8
Population: The Full Analysis Set with available data at Baseline. A mixed model for repeated measurements (MMRM) based on observed cases was used. "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 140 | 144
scores on a scale
  Week 1 (n=139, 142) | -1.02 (0.226) | -1.09 (0.228)
  Week 4 (n=130, 135) | -1.84 (0.273) | -2.28 (0.273)
  Week 8 (n=111, 124) | -2.55 (0.316) | -2.62 (0.308)

17. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Social Functioning Subscore at Other Weeks Assessed
Description: as for outcome 7
Time Frame: Baseline to Weeks 2 and 4
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 139 | 143
scores on a scale
  Week 2 (n=137, 143) | 11.96 (1.803) | 14.06 (1.820)
  Week 4 (n=129, 134) | 17.12 (1.993) | 16.22 (1.999)

18. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Physical Functioning Subscore at Each Week Assessed
Description: The Medical Outcomes Study SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The physical functioning subscale assesses limitations in physical activities because of health problems. The sub-score scale ranges from 0 (best) - 100 (worst). LS means were from a mixed model for repeated measurements (MMRM).
Time Frame: Baseline to Weeks 2, 4 and 8
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 139 | 143
scores on a scale
  Week 2 (n=137, 143) | 1.54 (1.322) | 3.69 (1.336)
  Week 4 (n=129, 134) | 4.76 (1.424) | 4.22 (1.432)
  Week 8 (n=113, 125) | 3.50 (1.640) | 4.18 (1.609)

19. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Role-Physical Subscore at Each Week Assessed
Description: The Medical Outcomes Study SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The role-physical subscale assesses limitations in usual role activities because of physical health problems. The sub-score scale ranges from 0 (best) - 100 (worst). LS means were from a mixed model for repeated measurements (MMRM).
Time Frame: Baseline to Weeks 2, 4 and 8
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 139 | 143
scores on a scale
  Week 2 (n=137, 143) | 5.03 (1.901) | 4.90 (1.906)
  Week 4 (n=129, 134) | 8.65 (1.966) | 5.19 (1.967)
  Week 8 (n=113, 125) | 10.02 (1.998) | 7.74 (1.953)

20. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Bodily Pain Subscore at Each Week Assessed
Description: The Medical Outcomes Study SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The bodily pain sub-score scale ranges from 0 (best) - 100 (worst). LS means were from a mixed model for repeated measurements (MMRM).
Time Frame: Baseline to Weeks 2, 4 and 8
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 139 | 143
scores on a scale
  Week 2 (n=137, 143) | 7.24 (1.743) | 6.49 (1.755)
  Week 4 (n=129, 134) | 9.81 (1.756) | 8.96 (1.761)
  Week 8 (n=113, 125) | 10.14 (1.965) | 8.58 (1.915)

21. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) General Health Subscore at Each Week Assessed
Description: The Medical Outcomes Study SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The general health sub-score scale ranges from 0 (best) - 100 (worst). LS means were from a mixed model for repeated measurements (MMRM).
Time Frame: Baseline to Weeks 2, 4 and 8
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 139 | 143
scores on a scale
  Week 2 (n=137, 143) | 2.79 (1.095) | 3.61 (1.109)
  Week 4 (n=129, 134) | 4.85 (1.204) | 1.76 (1.212)
  Week 8 (n=113, 125) | 6.14 (1.391) | 3.90 (1.365)

22. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Vitality Subscore at Each Week Assessed
Description: The Medical Outcomes Study SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The vitality sub-score assesses energy and fatigue, and ranges from 0 (best) - 100 (worst). LS means were from a mixed model for repeated measurements (MMRM).
Time Frame: Baseline to Weeks 2, 4 and 8
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 139 | 143
scores on a scale
  Week 2 (n=137, 143) | 8.91 (1.528) | 10.46 (1.555)
  Week 4 (n=129, 134) | 12.48 (1.655) | 12.67 (1.671)
  Week 8 (n=113, 125) | 16.06 (1.828) | 14.65 (1.805)

23. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Role-Emotional Subscore at Each Week Assessed
Description: The Medical Outcomes Study SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The role-emotional subscale assesses limitations in usual role activities because of emotional problems. The sub-score scale ranges from 0 (best) - 100 (worst). LS means were from a mixed model for repeated measurements (MMRM).
Time Frame: Baseline to Weeks 2, 4 and 8
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 139 | 143
scores on a scale
  Week 2 (n=137, 143) | 14.54 (2.028) | 13.25 (2.041)
  Week 4 (n=129, 134) | 16.00 (2.055) | 15.00 (2.063)
  Week 8 (n=113, 125) | 21.64 (2.202) | 19.01 (2.159)

24. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Mental Health Subscore at Each Week Assessed
Description: The Medical Outcomes Study SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The mental health sub-score assesses general mental health (psychological distress and well-being) and ranges from 0 (best) - 100 (worst). LS means were from a mixed model for repeated measurements (MMRM).
Time Frame: Baseline to Weeks 2, 4 and 8
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 139 | 143
scores on a scale
  Week 2 (n=137, 143) | 10.32 (1.455) | 11.72 (1.470)
  Week 4 (n=129, 134) | 12.58 (1.610) | 15.12 (1.617)
  Week 8 (n=113, 125) | 17.95 (1.716) | 16.91 (1.686)

25. Secondary Outcome: Health Care Resource Utilization as Assessed by the Health Economic Assessment Questionnaire
Description: Healthcare resource utilization was assessed by the Health Economic Assessment (HEA) questionnaire, which monitors the participants absenteeism from work, as well as resource use such as visits to a general practitioner, outpatient and inpatient services, hospitalization, medications, and other relevant services over the past 8 weeks.
Time Frame: Baseline and Week 8
Population: Full analysis set with available data at Baseline (139 and 136 patients) and at Week 8 (122 and 131 patients).
Measure: Number; unit: participants
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 139 | 136
participants
  Baseline: Any resource use | 30 | 30
  Baseline: Any hospitalization-related services | 1 | 0
  Baseline: Hospitalization related to anxiety | 0 | 0
  Baseline: Any sick leave | 8 | 10
  Baseline: Sick leave related to anxiety | 7 | 4
  Week 8: Any resource use | 22 | 19
  Week 8: Any hospitalization-related service | 0 | 1
  Week 8: Hospitalization related to anxiety | 0 | 0
  Week 8: Any sick leave | 4 | 6
  Week 8: Sick leave related to anxiety | 2 | 1

ADVERSE EVENTS:
Time Frame: Safety was assessed during the 8-week core treatment period and a 4-week follow-up period.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Vortioxetine 5 mg
Serious Adverse Events (participants affected / at risk) | 3/151 | 1/148
Other Adverse Events (participants affected / at risk) | 65/151 | 89/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=151) | Vortioxetine 5 mg (N=148)
Prostate infection (Infections and infestations) | 1 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=151) | Vortioxetine 5 mg (N=148)
Nausea (Gastrointestinal disorders) | 7 | 37
Dry mouth (Gastrointestinal disorders) | 5 | 12
Diarrhoea (Gastrointestinal disorders) | 7 | 8
Constipation (Gastrointestinal disorders) | 2 | 5
Dyspepsia (Gastrointestinal disorders) | 2 | 3
Vomiting (Gastrointestinal disorders) | 1 | 3
Irritability (General disorders) | 4 | 2
Fatigue (General disorders) | 3 | 3
Nasopharyngitis (Infections and infestations) | 6 | 8
Upper respiratory tract infection (Infections and infestations) | 5 | 3
Viral upper respiratory tract infection (Infections and infestations) | 5 | 4
Gastroenteritis viral (Infections and infestations) | 0 | 4
Overdose (Injury, poisoning and procedural complications) | 1 | 3
Blood pressure increased (Investigations) | 7 | 1
Increased appetite (Metabolism and nutrition disorders) | 2 | 5
Decreased appetite (Metabolism and nutrition disorders) | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Headache (Nervous system disorders) | 13 | 15
Dizziness (Nervous system disorders) | 5 | 12
Somnolence (Nervous system disorders) | 3 | 9
Sinus headache (Nervous system disorders) | 4 | 1
Memory impairment (Nervous system disorders) | 0 | 3
Tremor (Nervous system disorders) | 1 | 3
Insomnia (Psychiatric disorders) | 6 | 7
Abnormal dreams (Psychiatric disorders) | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Hot flush (Vascular disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.